CLINICAL TRIAL: NCT05113225
Title: Sperm Micro-swim up; a Novel Technique to Process and Select in the Same Dish:a Sibling-oocyte-split Design)
Brief Title: Sperm Micro-swim up Technique; Process and Select in the Same Dish: a Sibling-oocyte-split Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Fertility Center, Egypt (Other)
Collaborators: Hawaa Fertility Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2021-10-08; First posted 2021-11-09 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2021-10

CONDITIONS: Assisted Reproductive Technology; Infertility
Keywords: Sperm; micro-swim up; ICSI; Semen processing; density gradient
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Single group of patients will be recruited in the study and each patient's oocytes will be divided into two groups and each group of patients will be injected with sperm processed by normal DG or H pattern micro- swim up technique. The PVP was used to produce the H pattern (length of about 2 cm from one side of the plate to the middle of the disk, total volume 10 μL). A small amount of semen (3 μL) was placed on one side of the H, and some time was allowed for it to migrate to the other side where the sperm was then collected. The dishes were incubated for three minutes allowing sperm migration along the outer perimeter of the H. After the completion of sperm migration, the plate was turned before the upload to avoid the contamination of the injection pipette by the sample.The injection pipette was introduced into the H-ICSI™ and used to immobilize a single sperm by crushing the membrane of its tail.
Who Masked: Participant, Care Provider
Masking Description: the oocytes of each patient will be randomly divided before denudation and will be distributed in the ICSI dishes of different previously described PVP pattern and sperm processing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DG-ICSI (Active Comparator): Oocytes of this arm will be injected using sperm previously processed by DG method and located in the commonly used ICSI dishes with the common PVP microdroplets
  Interventions: Procedure: Micro-swim up technique
- H pattern-ICSI (Experimental): Oocytes of this arm will be injected using sperm that directly located in a specific H pattern PVP droplets in a commonly used ICSI dishes without pre-processing of the semen
  Interventions: Procedure: Micro-swim up technique

INTERVENTIONS:
Procedure: Micro-swim up technique — processing and selection of the sperm for ICSI in the same dish

SUMMARY:
A sibling-Oocyte-split design will be conducted on oocytes before denudation and divided into two groups : control group (MII oocytes will be injected using sperm processed by Density gradient method) and sample group ( MII oocytes will be injected by sperm processed using micro-swim up technique)

DETAILED DESCRIPTION:
In This study investigators compare a novel sperm processing and selection method which is (fast, cheap and safe) with the well known processing method of sperm "Density gradient (DG)"

The dishes will be prepared with droplets of handling medium for oocytes (droplet volume 10 μL), and an H pattern using PVP will be produced, finally, all the droplets will be overlaid with mineral oil.

Control group : Oocytes will be injected using sperm after processing with DG and will be selected from control PVP microdroplets

Sample group: Sperm will be directly loaded in specific ICSI dishes where is the PVP microdroplets is prepared on "H" Pattern and will be selected from the far point from the deposition point and will be injected into the oocytes from the sample group All injected MII oocytes from both groups will then be cultured, with each group demarcated in separate place in the culture dish then according to the randomisation embryo transfer will be selected from one of both groups then the quality of the embryos will be reported and the pregnancy rate

ELIGIBILITY:
Inclusion Criteria:

* The normal & high responders were selected according to :

  * age: 18 - 40 years
  * anti-Müllerian hormone (AMH): > 1.0 ng/ml
  * number of aspirated oocytes:more than or equal 8
  * BMI < 34

Exclusion Criteria:

* Age > 40 years;
* AMH < 1.0 ng/mL;
* aspirated oocytes < 8.
* severe male factor
* Testicular aspirated sperm

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Number of top quality embryos | 4 or 5 days after ICSI procedure day
  the number of best embryos in each arm in Day 4 or Day 5

SECONDARY OUTCOMES:
Early Cleavage rate | 2 days after ICSI procedure day
  The early cleavage rate of oocytes from overall injected oocytes
chemical pregnancy rate | 14 days after embryo transfer day
  the quantitative serum HCG level that indicates positive pregnancy test for cases from over all cases

CONTACTS AND LOCATIONS:
Overall Officials: Sahar SA Eissa, PHD, Study Director — research team leader; Engy EA Abdallah, MSC, Study Chair — investigator & researcher
Locations (1):
- Royal Fertility Center, Al Mansurah, Daqahlya, Egypt

IPD SHARING:
Plan to Share IPD: No
Study protocols and outcome